CLINICAL TRIAL: NCT01224223
Title: Myeloid Suppressors in Inflammation
Status: Completed | Type: Observational
Sponsor: University of South Florida (Other)
Responsible Party: Principal Investigator, Richard Lockey, principal investigator, University of South Florida
Other Study IDs: MYELOID
Record Dates: First submitted 2010-10-18; First posted 2010-10-19 (Estimated); Last update posted 2012-06-28 (Estimated); Status verified 2010-10

CONDITIONS: Asthma
Keywords: asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- acute asthma exaecerbtion patients: Patients experiencing acute exacerbation of their asthma
- chronic asthma group: Two groups are being enrolled. The first group is chronic asthma patients with FEV1 below 80% and FEV1/FVC ratio reduced by 5%

SUMMARY:
Myeloid-derived suppressor cells (MDSC) have been studied for their ability to suppress T cell responses in vivo and in vitro. As a result, MDSC can regulate cellular responses to chronic inflammatory conditions such as cancer, leading to the induction of tolerance and, ultimately, tumor escape from immune surveillance.

ELIGIBILITY:
Inclusion

1. Ages eligible for study: 18 to 60 years
2. Genders eligible for study: male and female
3. Signed and dated written informed consent is obtained prior to study blood draw.
4. Subjects being actively treated for chronic moderate to severe asthma based on National Heart Lung and Blood Institute guidelines (figure 1). Subjects must carry the diagnosis of asthma (made by a physician) for a minimum of six months.
5. Subjects within the first seven days of an acute asthma exacerbation, as determined by the referring physician.
6. Able to give informed consent.

Exclusion Criteria:

1. Use of systemic corticosteroids within the previous two weeks.
2. Pregnant and/or lactating females.
3. Current tobacco use.
4. Severe psychiatric illness.
5. Current illicit substance abuse or dependence and/or abuse of alcohol.
6. Current use of anti-microbial medications.
7. Primary or secondary immunodeficiency.
8. Any clinically significant uncontrolled medical condition that would put the patient's safety at risk.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Ages eligible for study: 18 to 60 years Genders eligible for study: male and female Signed and dated written informed consent is obtained prior to study blood draw.
  Subjects being actively treated for chronic moderate to severe asthma based on National Heart Lung and Blood Institute guidelines (figure 1). Subjects must carry the diagnosis of asthma (made by a physician) for a minimum of six months.
  Subjects within the first seven days of an acute asthma exacerbation, as determined by the referring physician.Able to give informed consent.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2010-10; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
To identify and characterize specific cell types (human dendritic cells, myeloid-derived suppressor cells and T lymphocytes) that are present in acute and chronic asthma. | one year from start of study

CONTACTS AND LOCATIONS:
Overall Officials: Richard Lockey, MD, Principal Investigator — USF Asthma, Allergy and Immunology CRU
Locations (1):
- USF Asthma, Allergy and Immunology CRU, Tampa, Florida, United States